CLINICAL TRIAL: NCT00655330
Title: A Prospective Randomized, Controlled, Open-labeled Trial of Probucol Combined With Valsartan in Patients With Diabetes Nephropathy
Brief Title: Probucol Combined With Valsartan in Reducing Proteinuria in Diabetes Nephropathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Wei Shi, Director of renal division of Guangdong General Hospital, Guangdong Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GPPH200603 -1
Record Dates: First submitted 2008-04-02; First posted 2008-04-09 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Type 2 Diabetes Mellitus; Nephropathy
Keywords: Type 2 diabetes mellitus; Nephropathy; valsartan; probucol; Proteinuria
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Kidney Diseases; Proteinuria | interventions — Valsartan; Probucol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Valsartan (160mg/day)is given in combination with Placebo
  Interventions: Drug: Valsartan; Drug: Placebo
- 2 (Experimental): Valsartan (160mg/day) + Probucol (750mg/day)
  Interventions: Drug: Valsartan; Drug: Probucol

INTERVENTIONS:
Drug: Valsartan — Valsartan (160mg/day)
Drug: Placebo — Placebo
  Arms: 1
Drug: Probucol — Probucol (750mg/day)
  Arms: 2

SUMMARY:
This is a prospective randomized controlled, open-labeled study to identify the efficacy of probucol in combination with valsartan in patients with Diabetes nephropathy. The reduction of urinary albumin or proteinuria will be the primary outcome studied. The expected study duration will be 48 weeks.

DETAILED DESCRIPTION:
a prospective randomized controlled, open-labeled study in patients with Diabetes nephropathy

* Arm 1: Valsartan + Probucol Valsartan (160mg/day) + Probucol (750mg/day)
* Arm 2: Valsartan + Placebo Valsartan (160mg/day) + Placebo

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes nephropathy
* Urinary albumin excretion 1-3g/24hours
* Serum creatinine < 3mg/dl

Exclusion Criteria:

* Type 1 diabetes mellitus
* Renal diseases other than type 2 Diabetes nephropathy
* Renal artery stenosis
* Severe heart diseases
* Tuberculosis

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2008-05; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
urinary albumin excretion or proteinuria at week 48 | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shi Wei, MD, PhD, Principal Investigator — Nephrology Dept.,Guangdong General Hospital
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China